CLINICAL TRIAL: NCT00834834
Title: Treating Suicidal Behavior and Self-Mutilation in Borderline Personality Disorder: Predictors of Change
Brief Title: Comparing Treatments for Self-Injury and Suicidal Behavior in People With Borderline Personality Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #5752/6777R; R01MH061017 (NIH); R01MH061017-06A2 (NIH)
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Borderline Personality Disorder; Suicide
Keywords: Suicidal and Self-Injurious Behavior
MeSH Terms: conditions — Borderline Personality Disorder; Suicide; Self-Injurious Behavior | interventions — Fluoxetine; Citalopram

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoxetine (Active Comparator): Participants will receive fluoxetine with clinical management, which may involve switching medication to citalopram, another SSRI.
  Interventions: Drug: Fluoxetine; Drug: Citalopram
- Dialectical behavior therapy (Active Comparator): Participants will receive dialectical behavioral therapy (DBT).
  Interventions: Behavioral: DBT

INTERVENTIONS:
Drug: Fluoxetine — Starting dose of 20 mg daily will increase over 4 weeks, depending on tolerability, up to 40 mg daily. Treatment will last 6 months.
  Other Names: Prozac
  Arms: Fluoxetine
Behavioral: DBT — One 60-minute individual therapy session and one 90-minute group therapy session every week. Treatment will last 6 months.
  Arms: Dialectical behavior therapy
Drug: Citalopram — Dose set by study psychiatrist, up to 60 mg daily. Treatment will last 6 months.
  Other Names: Celexa
  Arms: Fluoxetine

SUMMARY:
This study will compare the effectiveness of two treatments, dialectical behavior therapy versus fluoxetine with clinical management, for reducing the risk of self-injury and suicidal behavior in people with borderline personality disorder.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a chronic disorder in emotional regulation and is characterized by instability in self-image, mood, relationships, and behavior. People suffering from BPD have a high rate of self-injury and suicide attempts. This study will compare the effectiveness of two treatments for preventing self-injury and suicide in people with BPD: dialectical behavior therapy (DBT) and fluoxetine with clinical management. DBT is a behavioral therapy that teaches new coping skills to replace old strategies, including self-injury and attempted suicide. Fluoxetine is a selective serotonin reuptake inhibitor (SSRI) medication that has been used to treat BPD. Clinical management of fluoxetine, which is involved in administering the medication under normal conditions, refers to regular visits with a psychiatrist who will monitor medication effectiveness and side effects. Clinical management in this study may include adjusting the dosage of fluoxetine or prescribing a change in medication to citalopram, another SSRI.

Participation in this study will last 12 months, including all follow-up assessments. During the first study visit, participants will undergo baseline testing and be randomly assigned to receive either DBT or fluoxetine with clinical management. After a washout period, in which participants will transition off any medications they are currently taking, participants will receive 6 months of their assigned treatment. Participants receiving DBT will attend one 60-minute individual therapy session and one 90-minute group session every week. Participants assigned to the fluoxetine with clinical management condition will begin receiving 20 mg of fluoxetine daily and have their dose increased over the course of 4 weeks, based on tolerance, up to 40 mg. Participants assigned to fluoxetine may also be switched to citalopram, if the study psychiatrist thinks it will be more effective. Participants assigned to either fluoxetine or citalopram will undergo monthly blood tests to monitor the level of medication in their bodies.

Every 2 weeks, participants will undergo assessments of treatment effectiveness and side effects. After 2, 4, 6, 9, and 12 months, participants will undergo various neuropsychological tests and clinical interviews and self-report questionnaires about mood and life experiences. At study entry and at Weeks 12 and 24, participants will use a handheld computer to complete a week-long assessment of emotions. Fully healthy female participants will be asked to complete a functional magnetic resonance imaging (fMRI) scan, which will assess their ability to regulate emotions at the neural level. The fMRI scan and a stress test (for both men and women) will be performed at baseline and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual (DSM-IV) criteria for borderline personality disorder (BPD)
* Attempted suicide in the past 2 months
* At least one additional suicide attempt, suicide-related behavior, or self-injury episode in the past year
* Current suicidal ideation
* Able to be managed as an outpatient
* Not currently receiving optimum psychiatric treatment and agrees to notify study staff if any psychiatric care outside this study is sought. If care other than that permitted by the protocol is utilized, participants can no longer be enrolled in the study.
* Has a stable living arrangement at study entry
* Speaks English
* Willing and judged to be clinically able to undergo wash-out of psychotropic medications, except for occasional benzodiazepines use, for 2 to 6 weeks before treatment
* Females must be willing to use an effective method of birth control.

Exclusion Criteria:

* Meets the DSM-IV criteria for mental retardation or the following disorders: bipolar I, schizophrenia, delusional disorder, schizophreniform disorder, schizoaffective disorder, or psychotic disorder not otherwise specified (NOS)
* Needs priority treatment for acute medical illness or other debilitating problem, such as severe substance dependence or anorexia
* Pregnant
* Clinically too unstable to be maintained as an outpatient
* Has clearly failed adequate trials of fluoxetine and citalopram for a major depression in the past 2 years
* History of severe allergies, adverse drug reactions, or known allergy to fluoxetine or citalopram
* Clinically inadvisable for the participant to end current treatment
* Heart pacemaker body implant; other metal implants, such as shrapnel or surgical prostheses; or paramagnetic objects contained within the body, as assessed via a metal screening questionnaire, which may present a risk to the participant or interfere with the fMRI scan
* Diagnosed with Raynaud's disorder
* History of hypertension, cardiovascular disease, or abnormal electrocardiograms (EKGs)
* Claustrophobia or significant discomfort in enclosed space

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara H. Stanley, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment is from community clinicians, advertising and the emergency department.
Pre-assignment Details: All participants are washed out of psychotropic medications. Benzodiazapines are permitted for sleep.
Period: Overall Study
Arm/Group | Fluoxetine | Dialectical Behavior Therapy
Started | 42 | 42
Completed | 38 | 39
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine | Dialectical Behavior Therapy | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (7.8) | 30.6 (10.8) | 29.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 40 | 77
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 33 | 31 | 64
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Suicide Events
Description: Data on suicidal behavior was collected with the Columbia Suicide History Interview (CSHI), a semi-structured interview developed by our group. It is used to elicit history of the individual's actual suicide attempts , as well as specific questions concerning the circumstances surrounding any suicidal behavior and its degree of medical lethality. In addition to obtaining measurements of actual suicide attempts, the CSHI also captures suicide-related behaviors such as aborted and interrupted suicide attempts. An actual suicide attempt is operationally defined by the CSHI as a self-injurious act performed with at least some intent to die.
Time Frame: Measured after 6 months of treatment
Measure: Number; unit: suicide events
Arm/Group | Fluoxetine | Dialectical Behavior Therapy
Number analyzed (Participants) | 38 | 39
suicide events | 12 | 4

2. Secondary Outcome: Number of Participants With Suicide Events
Description: as for outcome 1
Time Frame: measured after 6 months of treatment
Measure: Number; unit: participants
Arm/Group | Fluoxetine | Dialectical Behavior Therapy
Number analyzed (Participants) | 38 | 39
participants | 6 | 4

ADVERSE EVENTS:
Time Frame: During 6 month treatment trial and 1 year follow up period.
Arm/Group | Fluoxetine | Dialectical Behavior Therapy
Serious Adverse Events (participants affected / at risk) | 14/38 | 5/39
Other Adverse Events (participants affected / at risk) | 0/38 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=38) | Dialectical Behavior Therapy (N=39)
Serious Adverse Event (Psychiatric disorders) | 14 (15) | 5 (8) — Includes suicidal behavior and psychiatric hospitalization Adverse Events were monitored/assessed without regard to the specific event and labeled as "Serious Adverse Event"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No